CLINICAL TRIAL: NCT05894408
Title: Portal Vein Occlusion is a Valuable Predictor for Postoperative Nausea and Vomiting in Patients With Liver Cancer: A Prospective Cohort Study
Brief Title: Portal Vein Occlusion is a Valuable Predictor for Postoperative Nausea and Vomiting
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SHDC22020204
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with portal vein occlusion
  Interventions: Other: this is no intervention
- patients without portal vein occlusion
  Interventions: Other: this is no intervention

INTERVENTIONS:
Other: this is no intervention — this is no intervention

SUMMARY:
Postoperative nausea and vomiting (PONV) is one of the most common and distressing postoperative complications. PONV risk assessment is recommanded to determine the number of medications or strategies for prophylaxis. Many well-known risk factors have been determined. However, no study has explored liver surgery-specific risk factors. This study aims to identify whether there was an association between portal vein occlusion and PONV among patients after liver surgery. Patients diagnosed with liver cancer and undergoing hepatectomy will be prospectively consecutively recruited. All enrolled patients receive PONV assessments within the first 24 postoperative hours. Logistic regression models will be used to investigate the effects of portal vein occlusion and the other variables on the occurrence of PONV in both univariate and multivariate analyses

DETAILED DESCRIPTION:
1. Design This is a single-centre, prospective cohort study performed at a tertiary teaching hospital in Shanghai, China.
2. Participants We calculated the sample size based on the rule-of-thumb method from logistic modelling as follows: a minimum of 10 events per predictor variable should be achieved based on simulation studies. The reported incidence of PONV among patients undergoing general surgery ranged from 30% to 50%. We used the lowest incidence of 30% to estimate the sample size. The expected variable number included in the logistic model was 9, and adjusting for a 10% of loss to follow-up, the sample size was 330.

   Patients will be prospectively consecutively recruited. Patients who are diagnosed with liver cancer and underwent hepatectomy are eligible. Inclusion criteria are age older than 18 years, planned admissions and elective surgery, and staying at least 24 hours in the surgical unit. We exclude patients with cognitive impairment and patients who had nausea and vomiting related to other existing diseases, such as gastroesophageal reflux disease. We also exclude patients who have severe postoperative complications, including massive abdominal hemorrhage, hepatic encephalopathy and portal vein thrombosis.
3. Setting The study will be conducted in the liver disease department in Zhongshan Hospital, Shanghai, China, which is the largest liver surgery department in eastern China. In 2018, the department performs nearly 3000 liver surgeries. The liver surgical department has 240 beds, and the department staff includes 106 nurses and physicians.
4. Data collection 4.1 Preoperative assessment All enrolled patients will receive preoperative assessments by trained investigators. The baseline demographic data and medical history will be recorded. We define smoking history as nicotine use before surgery, and history of motion sickness as nausea or vomiting when travelling in a car/boat/train/plane. Nonsmoking and history of motion sickness or PONV will be collected by interviewing patients and family members.

   4.2 Postoperative assessment All enrolled patients receive postoperative assessments by trained nurses. The use of postoperative opioids and the length of surgery are determined by checking the hospital information system to review surgery records and anaesthetic protocols within 24 hours after surgery. The time of portal vein occlusion will be recorded by the surgeon.
5. Surgery and postoperative management A standard general anaesthesia technique is used for all patients. Different operations are performed according to the preoperative conditions of each patient. S
6. Outcome measures Postoperative nausea and vomiting will be assessed hourly during the first two hours, every two hours for the following four hours and every four hours until the 24th hour by the first and the second authors to ensure high-quality data collection. PONV will be evaluated on a four-grade scale from 0 (no nausea and no vomiting), 1 (having nausea but no vomiting), 2 (having vomiting without stomach contents ) to 3 (having vomiting with stomach contents). A patient will be considered to have PONV if his or her PONV grade is 2 or more within the first 24 postoperative hours. PONV will be assessed by the first author, who is blinded to the result of portal vein occlusion.
7. Statistical analysis Statistical analyses are conducted using IBM-SPSS software version 22 (IBM Corp., Armonk, NY, USA), Empower (R) (www.empowerstats.com, X&Y solutions, Inc., Boston, MA), and R statistical software. Data are presented as the mean and standard deviation for continuous variables and as percentages for categorical variables. Normally distributed continuous variables are compared using one-way analysis of variance. The Pearson χ2 test is applied to all categorical variables. Logistic regression models are used to investigate the effects of portal vein occlusion and the other variables on the occurrence of PONV in both univariate and multivariate analyses. Independent variables are selected based on evidence from previous studies showing a significant relation to PONV and we also include other variables based on our clinical experience.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years, planned admissions and elective surgery, and staying at least 24 hours in the surgical unit

Exclusion Criteria:

* patients with cognitive impairment and patients who have nausea and vomiting related to other existing diseases, such as gastroesophageal reflux disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with liver cancer and underwent hepatectomy are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | up to 24 hours
  PONV will be evaluated on a four-grade scale from 0 (no nausea and no vomiting), 1 (having nausea but no vomiting), 2 (having vomiting without stomach contents ) to 3 (having vomiting with stomach contents).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Zhao WJ, Yu J, Zhou H, Shi Y, Gao J, Zhang Y. Duration of hepatic portal occlusion is a valuable predictor for postoperative nausea and vomiting in patients underwent liver resection for liver cancer. BMC Cancer. 2025 Jul 16;25(1):1177. doi: 10.1186/s12885-025-14592-0. PMID 40670918